CLINICAL TRIAL: NCT04975893
Title: A Phase 2, Non-Randomized, Long-Term Extension Study to Evaluate the Immunogenicity and Safety of Cytomegalovirus mRNA-1647 Vaccine Including a Booster Dose in a Subset of Participants Who Completed Study mRNA-1647-P202
Brief Title: A Long-Term Extension Study to Evaluate the Immunogenicity and Safety of Cytomegalovirus (CMV) mRNA-1647 Vaccine
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: ModernaTX, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: mRNA-1647-P202-EXT
Record Dates: First submitted 2021-07-09; First posted 2021-07-26 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Cytomegalovirus Infection
Keywords: Moderna; mRNA-1647; Cytomegalovirus; CMV; Cytomegalovirus Vaccine; Cytomegalovirus Infections; Cytomegalovirus Congenital; Virus Diseases; Infection Viral; DNA Virus Infections; Messenger RNA
MeSH Terms: conditions — Cytomegalovirus Infections; Virus Diseases; DNA Virus Infections | interventions — mRNA-1647 cytomegalovirus vaccine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Primary Extension Phase (Other): CMV-seropositive and CMV-seronegative participants who completed Study mRNA-1647-P202 will be followed every 6 months for 3 years in this study after the final visit in Study mRNA-1647-P202.
  Interventions: Biological: mRNA-1647
- Optional Booster Phase - BD Recipients (Experimental): Participants who opted to enroll into the optional Booster Phase will receive a single mRNA-1647 vaccine dose.
  Interventions: Other: mRNA-1647
- Optional Booster Phase - Observational Group (Other): Participants who opted to enroll into the Observational Group will be followed in the optional BP until BP Month 12.
  Interventions: Biological: mRNA-1647

INTERVENTIONS:
Biological: mRNA-1647 — No investigational product will be administered during the Primary Extension Phase or to the participants in the Observational Group.
  Arms: Optional Booster Phase - Observational Group; Primary Extension Phase
Other: mRNA-1647 — Lyophilized product that is reconstituted with saline then diluted with a special diluent to reach the desired concentration
  Arms: Optional Booster Phase - BD Recipients

SUMMARY:
The main purpose of the extension phase of this study is to evaluate the longer-term immune persistence of mRNA-1647 vaccine administered to CMV-seronegative and CMV-seropositive adults who completed Study mRNA-1647-P202 (NCT04232280). For participants in the optional booster phase (BP), the main purpose is to evaluate the long-term immunogenicity and safety of the mRNA-1647 vaccine in both participants receiving a booster dose (BD) and those not receiving a BD, and to additionally evaluate the reactogenicity in participants receiving a BD.

DETAILED DESCRIPTION:
The study aims to explore the long-term potential differences in immunogenicity and key safety parameters following mRNA-1647 administration, participants who completed study mRNA-1647-P202, who are CMV-seronegative and who did not seroconvert due to primary CMV infection during the study will be enrolled. Study mRNA-1647-P202 participants who were CMV-seropositive at baseline, randomized to receive mRNA-1647 injection, and completed their final study visit will also be enrolled.

No study treatment will be administered during the primary extension phase of this study. Eligible participants enrolling in the primary extension phase who completed Study mRNA-1647-P202 may have received mRNA-1647 (either low dose, medium dose, or high dose) or placebo in CMV-seronegative participants and mRNA-1647 (either low dose, medium dose, or high dose) in CMV-seropositive participants.

In the optional BP, consenting and eligible participants will receive a single BD of the mRNA-1647 vaccine (medium dose). In the Observational Group of the optional BP, consenting and eligible participants will not receive study treatment.

ELIGIBILITY:
Inclusion Criteria:

Primary Extension Phase:

* Male and female participants who were CMV-seronegative at the Study mRNA-1647-P202 Screening visit, completed the final Study mRNA-1647-P202 visit, and remained CMV-seronegative at Screening for Study mRNA-1647-P202-EXT.
* Male and female participants who were CMV-seropositive at the Study mRNA-1647-P202 Screening visit, were randomized to receive mRNA-1647 injection (and not placebo), and completed the final visit in Study mRNA-1647-P202.
* Understands and agrees to comply with the trial procedures and provides written informed consent.
* According to the assessment of the Investigator, is in good general health and is capable of complying with trial procedures.

Optional Booster Phase:

For BD Recipients:

- CMV-seronegative and CMV-seropositive participants who received mRNA-1647 medium dose injection (and not placebo or other dose levels) in Study mRNA-1647-P202, including participants who enrolled in the Primary Extension Phase of Study mRNA-1647-P202-EXT and participants who were eligible but did not previously enroll in the Primary Extension Phase of Study mRNA-1647-P202-EXT are eligible to receive a BD in the optional BP.

For Observational Group:

- CMV-seronegative and CMV-seropositive participants who received mRNA-1647 low dose or high dose injection (and not placebo or mRNA-1647 medium dose injection) in Study mRNA-1647-P202, including participants who enrolled in the Primary Extension Phase of Study mRNA-1647-P202-EXT and participants who were eligible but did not previously enroll in the Primary Extension Phase of Study mRNA-1647-P202-EXT are eligible to enroll in the observational group.

Exclusion Criteria:

Primary Extension Phase:

* Receipt of any CMV vaccine other than mRNA-1647.
* Diagnosis or condition that, in the judgment of the Investigator, may affect participant safety, assessment of safety endpoints, assessment of immune response, or adherence to trial procedures, including any medical, psychiatric, or occupational condition that, in the opinion of the Investigator, might pose additional risk due to participation in the study or could interfere with the interpretation of study results.

Optional Booster Phase:

For BD Recipients:

- Participants from the placebo, mRNA-1647 low dose, or mRNA-1647 medium dose groups in Study mRNA-1647-P202.

For Observational Group:

- Participants from the placebo or mRNA-1647 medium dose groups in study mRNA-1647-P202.

Note: Other protocol-defined inclusion/exclusion criteria apply

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 135 (Actual)
Dates: Start 2021-06-18 (Actual); Primary Completion 2026-01-19 (Actual); Study Completion 2026-01-19 (Actual)

PRIMARY OUTCOMES:
Primary Extension Phase: Geometric Mean Titers (GMTs) of Antigen-Specific Neutralizing Antibody (nAb) and Binding Antibody (bAb) | Up to 3 years
BP: GMTs of Antigen-Specific nAb and bAb | BP Month 0, BP Month 1, BP Month 3, BP Month 6, and BP Month 12
BP: Number of Participants with Solicited Adverse Reactions (ARs) | Up to BP Day 7 (7 days after BP vaccination)
BP: Number of Participants with Unsolicited Adverse Events (AEs) | Up to BP Day 28 (28 days after BP vaccination)
BP: Number of Participants with Medically-Attended AEs (MAAEs) | Up to BP Month 6 (6 months after BP vaccination)
BP: Number of Participants with Adverse Events of Special Interest (AESIs), Serious Adverse Events (SAEs), and AEs Leading to Discontinuation of Study | Up to BP Month 12

SECONDARY OUTCOMES:
Primary Extension Phase: Number of Participants With AEs Leading to Study Discontinuation | Up to 3 years
Primary Extension Phase: Number of Participants With SAEs | Up to 3 years

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - Optimal Research, LLC, Peoria, Illinois
  - Johnson County Clin-Trials, Inc., Lenexa, Kansas
  - Alliance for Multispeciality Research, LLC, Lexington, Kentucky
  - Tekton Research Inc, Austin, Texas
  - Crossroads Clinical Research (Victoria), Victoria, Texas
  - J. Lewis Research, Inc. / Foothill Family Clinic South, Salt Lake City, Utah